CLINICAL TRIAL: NCT02115789
Title: Perceptions of Aesthetic Outcomes of Zigzag and Linear Scars
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 346072
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Linear Scar; Zigzag Scar
Keywords: cicatrix; Demonstrate; that there; is no perception of superiority
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Survey Group: Adult male or female volunteers.
  Interventions: Behavioral: Visual Analog Scale

INTERVENTIONS:
Behavioral: Visual Analog Scale — Subjects will review examples of both linear and zigzag scars and rate the aesthetic appearance of both configurations of scars on a scale of 1 through 10, with 1 being "normal skin" and 10 being "the worst scar imaginable".

SUMMARY:
Surgical wounds can be closed in several manners. Some physicians believe that closure in a straight line produces a scar that is more visible and slightly raised when compared to closure in a zigzagging fashion. The researchers of this study believe that there is no difference in the cosmetic appearance of one type of wound closure over the other. To evaluate this, they will provide a survey with visual aids to volunteers to rate the appearance of a straight line scar versus a zigzag scar.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 years or older

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the dermatology clinic at UC Davis Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 876 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Subjects will review examples of both linear and zigzag scars and rate the aesthetic appearance of both configurations of scars on a scale of 1 through 10, with 1 being "normal skin" and 10 being "the worst scar imaginable". | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, M.D., Principal Investigator — University of California, Davis
Locations (1):
- UC Davis, Department of Dermatology, Sacramento, California, United States

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical